CLINICAL TRIAL: NCT06387953
Title: Mitigation of Emergence Agitation Through Implementation of Masimo Bridge Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor of the study and the University of Washington were not able to come to an agreement on the intellectual property provisions. Therefore, this study will not be carried out.
Sponsor: University of Washington (Other)
Responsible Party: Principal Investigator, Jeffrey Kirsch, Professor: Anesthesiology and Pain Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: STUDY00019480
Record Dates: First submitted 2024-03-30; First posted 2024-04-29 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Emergence Delirium; Agitation, Emergence
MeSH Terms: conditions — Emergence Delirium | interventions — Bridge Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Bridge Therapy (Active Comparator): Subjects receive the Bridge therapy
  Interventions: Device: Bridge Therapy
- Placebo (Placebo Comparator): Subjects receive a placebo or sham therapy
  Interventions: Device: Sham Therapy

INTERVENTIONS:
Device: Bridge Therapy — After the patient has been intubated in the operating room - the Bridge device intervention will be applied to the subject's ear by a trained study team member. At the time of the pre-incision pause, Initiation of the intervention (Bridge therapy) will begin and will be continued throughout the surgery. The intervention will continue for 24 hours after extubation.
  Arms: Bridge Therapy
Device: Sham Therapy — After the patient has been intubated in the operating room - the Bridge device intervention will be applied to the subject's ear by a trained study team member. At the time of the pre-incision pause, Initiation of the intervention (Sham therapy) will begin and will be continued throughout the surgery. The intervention will continue for 24 hours after extubation.
  Arms: Placebo

SUMMARY:
This is a randomized, prospective, double-blinded (patient and outcome-assessor) trial. Our goal is to assess efficacy of Bridge Therapy (versus sham bridge therapy) to prevent emergence agitation following general anesthesia.

Primary Objective: Activation of Bridge Therapy from the time of the pre incision "time out" until 24 hours after admission to the PACU (Post Anesthesia Care Unit) is associated with reduced frequency and intensity of emergence agitation.

Secondary Objective: Bridge Therapy activation will also result in a lower incidence of rescue pharmacologic treatment of agitation.

Tertiary Objective: Activation of Bridge Therapy during a stable anesthetic state is associated with a reduced Patient State Index as measured on Sedline

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-90
2. English Speaking
3. ASA Physical Status between I-IV
4. Undergoing a surgical procedure at HMC
5. Patient answers "yes" to one of the following below:

   1. Do you drink 7 or more alcoholic beverages per week?
   2. Do you use (smoke or eat) cannabis (or other recreational drugs) on a weekly basis?
   3. Have you felt disoriented, aggressive, angry, or delirious after waking up from a previous surgery?
   4. Have you been told by a care provider or friend/family member that you woke up from surgery in the past disoriented, confused, or aggressive/angry?
   5. Have you been diagnosed with post-traumatic stress disorder (PTSD)?

Exclusion Criteria:

1. <18 years old, >90 years old
2. Intubated patients
3. Pregnant by HMC lab test
4. Non-English Speaking
5. Has a cardiac pacemaker
6. Hx of bleeding condition
7. Skin issues where the device would be applied, this includes: Dermatitis, Psoriasis vulgaris, skin breakdown, skin integrity compromised.
8. Plan to use dexmedetomidine as part of the anesthetic technique
9. Plan to use sedline for clinical anesthetic management during operating procedure.
10. Patients with previous history of sensitivity to compound benzoin tincture.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-08-27 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Emergence agitation | From time of the pre incision "time out" until 24 hours after admission to the PACU (Post-Anesthesia Care Unit)
  Frequency of emergence agitation following general anesthesia will be collected every 15 minutes in the PACU. Once discharged from the PACU this will be measured every 12 hours.
Emergence agitation | time out" until 24 hours after admission to the PACU (Post-Anesthesia Care Unit)
  Intensity of emergence agitation following general anesthesia will be measured by the Riker Sedation Agitation Scale (RSAS). The maximum score is 7, the minimum score is 1.
  A high scores means a worse outcome (higher agitation).

SECONDARY OUTCOMES:
Rescue pharmacologic treatment of agitation | From time of the pre incision "time out" until 24 hours after admission to the PACU (Post-Anesthesia Care Unit)
  Incidence of rescue pharmacologic treatment of agitation following general anesthesia. This will be measured by the number of times rescue pharmacological treatment was given.

OTHER OUTCOMES:
Patient State Index | From time of the pre incision "time out" until 24 hours after admission to the PACU (Post-Anesthesia Care Unit)
  Patient State Index or PSI is a clinically validated measure of the effect of anesthesia and sedation. PSI is measured on a Sedline Sedation Monitor. PSI values range from 0 (total cortical silence) to 100 (awake state), and 25-50 indicates the optimal hypnotic state for surgical anesthesia.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Kirsch, MD, Principal Investigator — University of Washington

IPD SHARING:
Plan to Share IPD: No